CLINICAL TRIAL: NCT01007552
Title: A Multicenter Phase II Study of Gemcitabine, Capecitabine and Bevacizumab for Locally Advanced or Metastatic Adenocarcinoma of the Gall Bladder or Biliary Ducts.
Brief Title: A Study of Gemcitabine, Capecitabine and Bevacizumab to Treat Cancer of the Gall Bladder or Bile Ducts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 150509
Record Dates: First submitted 2009-11-02; First posted 2009-11-04 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Cholangiocarcinoma
Keywords: Biliary Duct Cancer; Cancer of the Gallbladder; Adenocarcinoma of the Gall Bladder; Adenocarcinoma of the Biliary Ducts; Cholangiocarcinoma; Extrahepatic cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Gemcitabine; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Capecitabine and Bevacizumab (Experimental): Estimate the toxicity of the regimen, and estimate the quality of life (QOL).
  Interventions: Drug: Gemcitabine, Capecitabine and Bevacizumab

INTERVENTIONS:
Drug: Gemcitabine, Capecitabine and Bevacizumab — Bevacizumab 15 mg/ kg every 3 weeks, starting day 1; Capecitabine 650 mg/m2 bid x 14 days starting day 1, Gemcitabine 1000 mg/m2 days 1 and 8, cycles to be repeated every 21 days.

SUMMARY:
To assess the proposed therapy for patients with advanced gallbladder or biliary cancers.

DETAILED DESCRIPTION:
The primary objective of this study is to assess progression free survival with proposed therapy for patients with locally advanced or metastatic adenocarcinoma of the gallbladder or biliary ducts.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed gallbladder or biliary tract adenocarcinoma that is unresectable or metastatic, or metastatic adenocarcinoma which is radiologically confirmed to be of gallbladder or biliary origin. No prior systemic therapy for metastatic disease. Prior adjuvant therapy is permitted if completed over 6months ago.
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of bevacizumab in combination with gemcitabine in patients over 18 years of age, children are excluded from this study, but will be eligible for future pediatric phase 1 combination trials.
* ECOG performance status 0 or 1.
* Life expectancy > 3 months.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥ 3,000/microL
  * absolute neutrophil count ≥ 1,500/microL
  * platelets ≥ 1OO,OOO/microL
  * total bilirubin ≤ 2 mg/dl
  * AST or ALT ≤ 5 times upper limit of normal (UNL) for subjects with documented liver metastases; ≤ 2.5 times UNL for subjects without evidence of liver metastases.
  * creatinine < 1.5 mg/dL or 24 hour urine creatinine clearance > 50 ml/min.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Signed, written informed consent document.
* Patient must have measurable disease

Exclusion Criteria:

* Subjects meeting any of the following criteria are ineligible for study entry:
* Compromised renal or hepatic function.
* Screening clinical laboratory values INR ≥ 1.5 (except those subjects who are receiving full-dose warfarin)
* Hemoglobin < 9 gm/dL (may be transfused or receive epoetin alfa (e.g., Epogen@) to maintain or exceed this level).
* Bevacizumab risk factors: History of serious systemic disease, including uncontrolled hypertension (blood pressure of greater than 160/110 mmHg on medication), prior history of hypertensive crisis or hypertensive encephalopathy, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), or clinically significant peripheral vascular disease (Grade II or greater).
* Presence of central nervous system or brain metastases.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study; fine needle aspirations or core biopsies within 7 days prior to Day O.
* Pregnancy (positive pregnancy test) or lactation.
* 24 hour urine creatinine clearance < 50 ml/min or urine protein/creatinine ratio greater than or equal to 1.0 at screening.
* Serious, nonhealing wound, ulcer, or bone fracture.
* Evidence of bleeding diathesis or coagu1opathy.
* Recent (less than or equal to six months) arterial thromboembolic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, or myocardial infarction (MI).
* Inability to comply with study and/or follow-up procedures.
* Patients with known duodenal or gastric wall involvement should be excluded.
* Patients with suspected involvement of stomach or duodenum should have screening endoscopies to exclude the same prior to therapy.
* Patients with esophageal or gastric varices.
* Patients with recent hemoptysis (within 1 week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine, Capecitabine and Bevacizumab
Started | 50
Completed | 49
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Gemcitabine, Capecitabine and Bevacizumab
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Study is to Assess Progression Free Survival (PFS) With Proposed Therapy for Patients With Locally Advanced or Metastatic Gallbladder and Biliary Cancers.
Description: Progression will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST 1.0). Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria. Note: Lesions are either measurable or non-measurable using the criteria provided below. The term "evaluable" in reference to measurability will not be used because it does not provide additional meaning or accuracy.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Capecitabine and Bevacizumab
Number analyzed (Participants) | 50
months | 8.1 [5.3 to 9.9]

2. Secondary Outcome: Estimate the Proportion of Patients With Clinical Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: as for outcome 1
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine, Capecitabine and Bevacizumab
Number analyzed (Participants) | 50
percentage of participants | 24 [13 to 38]

3. Secondary Outcome: Assess the Toxicity of the Regimen.
Description: Number of patients with Serious Adverse Events. Please refer to the adverse event reporting for more detail.
Time Frame: up to 5 years
Population: All treated and eligible patients
Measure: Number; unit: participants
Arm/Group | Gemcitabine, Capecitabine and Bevacizumab
Number analyzed (Participants) | 50
participants | 30

4. Secondary Outcome: Assess the Change in the Quality of Life Among Patients Using the FACT-Hep (Version 4) for Hepatobiliary Cancers.
Description: We utilized the FACT-HEP TOTAL SCORE (version 4) quality-of-life scale, which is a 45 item scale ranging from 96-178. Higher scores of the reflect better quality of life.
  For a Detailed description see:
  Nancy Heffernan, David Cella, Kimberly Webster, Linda Odom, Mary Martone, Steven Passik, Marilyn Bookbinder, Yuman Fong, William Jarnagin, and Leslie Blumgart: Measuring Health-Related Quality of Life in Patients With Hepatobiliary Cancers: The Functional Assessment of Cancer Therapy-Hepatobiliary Questionnaire. Journal of Clinical Oncology, Vol 20, No 9 (May 1), 2002: pp 2229-2239.
  No subscales were analyzed.
  .
Time Frame: Baseline, Day 22 and Day 43
Population: All treated and eligible patients. Some measures were not complete for leading to missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gemcitabine, Capecitabine and Bevacizumab
Number analyzed (Participants) | 49
units on a scale
  Baseline | 136.7 (20.8)
  Cycle 2 | 135.6 (22.1)
  Cycle 3 | 139.9 (16.7)

5. Secondary Outcome: Assess Overall Survival (OS)
Time Frame: as for outcome 1
Population: All treated and eligible patients
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Capecitabine and Bevacizumab
Number analyzed (Participants) | 50
months | 10.2 [7.5 to 13.7]

6. Secondary Outcome: Circulating Tumor Cells (CTC) Will be Assessed at Baseline, Day 22 and Day 43
Description: Mean number of CTCs in 7.5 ml of whole blood
Time Frame: baseline, day 22 and day 43
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Gemcitabine, Capecitabine and Bevacizumab
Number analyzed (Participants) | 50
cells
  Baseline | 2.3 (0.9)
  Day 22 | 1.0 (0.4)
  Day 43 | 0.8 (0.7)

7. Secondary Outcome: Collect Samples at Baseline, Day 8 and Day 43 for Future Biomarker Studies and Development of Profiles of Responders to Anti-VEGF Therapy (Optional)
Description: This was a tissue banking end point of sample collection for future studies. No analysis was completed.
Time Frame: Baseline, day 8 and day 43
Population: No patients were analyzed and no data were collected for this Outcome Measure. This was an optional aim and the research team decided to opted out of analyzing.
Arm/Group | Gemcitabine, Capecitabine and Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Gemcitabine, Capecitabine and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 30/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Capecitabine and Bevacizumab (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 (3)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3)
Pericarditis (Cardiac disorders) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (12)
Colitis (Gastrointestinal disorders) | 3 (9)
Constipation (Gastrointestinal disorders) | 1 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (6)
Intestinal obstruction (Gastrointestinal disorders) | 2 (6)
Large intestine perforation (Gastrointestinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 2 (6)
Varices oesophageal (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 2 (6)
Fatigue (General disorders) | 2 (6)
Pyrexia (General disorders) | 4 (12)
Cholangitis (Hepatobiliary disorders) | 4 (15)
Cholecystitis (Hepatobiliary disorders) | 1 (3)
Hepatic failure (Hepatobiliary disorders) | 1 (6)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (3)
Abdominal infection (Infections and infestations) | 1 (3)
Bacteraemia (Infections and infestations) | 3 (12)
Biliary sepsis (Infections and infestations) | 1 (6)
Clostridium difficile colitis (Infections and infestations) | 1 (3)
Kidney infection (Infections and infestations) | 1 (3)
Liver abscess (Infections and infestations) | 1 (3)
Pneumonia (Infections and infestations) | 1 (6)
Sepsis (Infections and infestations) | 3 (9)
Kidney injury molecule-1 (Investigations) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (6)
Cerebrovascular accident (Nervous system disorders) | 1 (3)
Mental impairment (Nervous system disorders) | 1 (3)
Confusional state (Psychiatric disorders) | 1 (3)
Renal failure (Renal and urinary disorders) | 2 (6)
Renal failure acute (Renal and urinary disorders) | 1 (3)
Urethral stenosis (Renal and urinary disorders) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Deep vein thrombosis (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 1 (3)
Vascular occlusion (Vascular disorders) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Capecitabine and Bevacizumab (N=50)
Anaemia (Blood and lymphatic system disorders) | 34 (399)
Leukopenia (Blood and lymphatic system disorders) | 38 (837)
Lymphopenia (Blood and lymphatic system disorders) | 34 (369)
Neutropenia (Blood and lymphatic system disorders) | 29 (522)
Thrombocytopenia (Blood and lymphatic system disorders) | 31 (435)
Pericardial effusion (Cardiac disorders) | 2 (6)
Tachycardia (Cardiac disorders) | 1 (3)
Ear pain (Ear and labyrinth disorders) | 1 (3)
Vertigo (Ear and labyrinth disorders) | 1 (3)
Abnormal sensation in eye (Eye disorders) | 1 (3)
Cataract (Eye disorders) | 1 (3)
Dacryostenosis acquired (Eye disorders) | 1 (3)
Dry eye (Eye disorders) | 1 (3)
Eye haemorrhage (Eye disorders) | 1 (6)
Keratitis (Eye disorders) | 1 (3)
Periorbital oedema (Eye disorders) | 1 (3)
Photophobia (Eye disorders) | 2 (6)
Vision blurred (Eye disorders) | 6 (21)
Vitreous floaters (Eye disorders) | 1 (3)
Abdominal discomfort (Gastrointestinal disorders) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 10 (36)
Abdominal pain (Gastrointestinal disorders) | 20 (84)
Abdominal pain lower (Gastrointestinal disorders) | 2 (9)
Abdominal pain upper (Gastrointestinal disorders) | 5 (21)
Anal fissure (Gastrointestinal disorders) | 1 (6)
Anal haemorrhage (Gastrointestinal disorders) | 1 (3)
Ascites (Gastrointestinal disorders) | 9 (54)
Cheilitis (Gastrointestinal disorders) | 1 (3)
Colitis (Gastrointestinal disorders) | 1 (6)
Constipation (Gastrointestinal disorders) | 24 (129)
Diarrhoea (Gastrointestinal disorders) | 23 (273)
Dry mouth (Gastrointestinal disorders) | 8 (24)
Dyspepsia (Gastrointestinal disorders) | 10 (36)
Faecal incontinence (Gastrointestinal disorders) | 1 (3)
Flatulence (Gastrointestinal disorders) | 4 (27)
Gingival bleeding (Gastrointestinal disorders) | 1 (3)
Glossodynia (Gastrointestinal disorders) | 1 (3)
Haematochezia (Gastrointestinal disorders) | 3 (9)
Intestinal perforation (Gastrointestinal disorders) | 1 (3)
Loose tooth (Gastrointestinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 31 (378)
Stomatitis (Gastrointestinal disorders) | 17 (84)
Vomiting (Gastrointestinal disorders) | 22 (210)
Asthenia (General disorders) | 7 (27)
Chest pain (General disorders) | 3 (9)
Chills (General disorders) | 17 (126)
Fatigue (General disorders) | 40 (362)
Gait disturbance (General disorders) | 2 (6)
Generalised oedema (General disorders) | 1 (6)
Influenza like illness (General disorders) | 5 (18)
Injection site rash (General disorders) | 1 (3)
Localised oedema (General disorders) | 2 (6)
Mucosal inflammation (General disorders) | 12 (84)
Non-cardiac chest pain (General disorders) | 2 (9)
Oedema (General disorders) | 4 (21)
Oedema peripheral (General disorders) | 24 (129)
Pain (General disorders) | 3 (12)
Pyrexia (General disorders) | 19 (243)
Hyperbilirubinaemia (Hepatobiliary disorders) | 19 (144)
Bacteraemia (Infections and infestations) | 1 (3)
Bacterial infection (Infections and infestations) | 1 (3)
Bronchitis (Infections and infestations) | 1 (3)
Candidiasis (Infections and infestations) | 1 (3)
Cellulitis (Infections and infestations) | 5 (24)
Fungal infection (Infections and infestations) | 1 (3)
Gingival infection (Infections and infestations) | 1 (3)
Infection (Infections and infestations) | 5 (15)
Laryngitis (Infections and infestations) | 1 (3)
Liver abscess (Infections and infestations) | 1 (3)
Nasopharyngitis (Infections and infestations) | 1 (3)
Pneumonia (Infections and infestations) | 1 (3)
Pneumonia klebsiella (Infections and infestations) | 1 (3)
Rhinitis (Infections and infestations) | 3 (9)
Sinusitis (Infections and infestations) | 2 (6)
Tooth abscess (Infections and infestations) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (6)
Urinary tract infection (Infections and infestations) | 6 (18)
Contusion (Injury, poisoning and procedural complications) | 3 (9)
Fall (Injury, poisoning and procedural complications) | 2 (9)
Joint injury (Injury, poisoning and procedural complications) | 1 (3)
Alanine aminotransferase increased (Investigations) | 32 (363)
Aspartate aminotransferase increased (Investigations) | 34 (369)
Blood albumin decreased (Investigations) | 1 (6)
Blood alkaline phosphatase (Investigations) | 1 (3)
Blood alkaline phosphatase increased (Investigations) | 22 (153)
Blood amylase increased (Investigations) | 1 (3)
Blood bilirubin increased (Investigations) | 1 (3)
Blood calcium decreased (Investigations) | 1 (3)
Blood creatinine increased (Investigations) | 15 (117)
Blood potassium decreased (Investigations) | 1 (6)
Blood urea increased (Investigations) | 1 (3)
Heart rate irregular (Investigations) | 1 (3)
International normalised ratio increased (Investigations) | 5 (39)
Neutrophil count decreased (Investigations) | 2 (9)
Platelet count decreased (Investigations) | 1 (3)
Troponin I increased (Investigations) | 1 (3)
Weight decreased (Investigations) | 14 (60)
Weight increased (Investigations) | 2 (9)
White blood cell count decreased (Investigations) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 23 (105)
Dehydration (Metabolism and nutrition disorders) | 5 (15)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 2 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 19 (345)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (48)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 33 (399)
Hypocalcaemia (Metabolism and nutrition disorders) | 22 (165)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 17 (93)
Hyponatraemia (Metabolism and nutrition disorders) | 34 (303)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (66)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (30)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (15)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 (60)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (24)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (6)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3)
Dizziness (Nervous system disorders) | 18 (54)
Dysgeusia (Nervous system disorders) | 18 (81)
Headache (Nervous system disorders) | 16 (72)
Hypoaesthesia (Nervous system disorders) | 5 (21)
Leukoencephalopathy (Nervous system disorders) | 1 (3)
Neuropathy peripheral (Nervous system disorders) | 9 (33)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (12)
Restless legs syndrome (Nervous system disorders) | 1 (3)
Sinus headache (Nervous system disorders) | 4 (21)
Somnolence (Nervous system disorders) | 2 (6)
Tardive dyskinesia (Nervous system disorders) | 1 (3)
Anxiety (Psychiatric disorders) | 10 (36)
Confusional state (Psychiatric disorders) | 3 (15)
Depression (Psychiatric disorders) | 14 (66)
Hallucination (Psychiatric disorders) | 1 (6)
Insomnia (Psychiatric disorders) | 14 (57)
Mental status changes (Psychiatric disorders) | 3 (9)
Bladder spasm (Renal and urinary disorders) | 1 (3)
Haematuria (Renal and urinary disorders) | 1 (3)
Micturition urgency (Renal and urinary disorders) | 1 (3)
Pollakiuria (Renal and urinary disorders) | 1 (3)
Proteinuria (Renal and urinary disorders) | 3 (48)
Urinary retention (Renal and urinary disorders) | 2 (9)
Pelvic pain (Reproductive system and breast disorders) | 1 (12)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (45)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 (126)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (78)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (24)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (21)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (12)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (15)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (18)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (21)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (9)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (30)
Erythema (Skin and subcutaneous tissue disorders) | 3 (9)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (27)
Nail disorder (Skin and subcutaneous tissue disorders) | 7 (21)
Night sweats (Skin and subcutaneous tissue disorders) | 8 (30)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 25 (132)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (42)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 12 (69)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 12 (36)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (3)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 (3)
Cataract operation (Surgical and medical procedures) | 1 (3)
Sinus operation (Surgical and medical procedures) | 1 (3)
Deep vein thrombosis (Vascular disorders) | 2 (9)
Embolism arterial (Vascular disorders) | 1 (3)
Flushing (Vascular disorders) | 1 (3)
Haematoma (Vascular disorders) | 1 (3)
Hot flush (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 14 (90)
Hypotension (Vascular disorders) | 6 (21)
Thrombosis (Vascular disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes